CLINICAL TRIAL: NCT02587741
Title: Comparison of Diabetes Retinopathy Among Type 2 Diabetic Patients Treated With Different Regimens: a Multicentre Randomized Parallel-group Clinical Trial
Brief Title: Comparison of Diabetes Retinopathy Among Type 2 Diabetic Patients Treated With Different Regimens
Acronym: CORRECT
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yanming Chen, Professor of Internal Medicine, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Third SunYetSan
Record Dates: First submitted 2015-10-18; First posted 2015-10-27 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Diabetic Retinopathy
Keywords: type 2 diabetes mellitus; Diabetic Retinopathy; glucose fluctuation; oxidative stress; Insulin; Oral drugs
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Metformin; Acarbose; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- oral drugs (Experimental): oral anti-diabetic drugs only.metformin,start from 500mg bid,if blood glucose dose not reach the standard，added to 500mg tid→1000mg bid.if metformin reach the biggest dosage，added gliclazide modified release tablets，from 30mg qd,if blood glucose dose not reach the standard,add dosage 30mg qd→60 mg qd→90mg qd→120mg qd(max).if still not reach the target，add acarbose 50mg tid
  Interventions: Drug: Metformin
- lantus (Experimental): basal insulin combine with oral drugs,started with insulin glargine 0.2 u/kg subcutaneous injection at 10pm（at 8am if patients are night workers）,add dosage if glucose dose not reach the target.after that,you can add oral drugs ,as Group Oral Drugs.
  Interventions: Drug: Lantus
- Novomix30 (Experimental): premixed insulin combine with oral drugs,started with premixed insulin subcutaneous injection(0.4-0.6 u/kg divided into half before breakfast and dinner),and add dosage if glucose dose not reach the target.after that,you can add oral drugs ,as Group Oral Drugs .
  Interventions: Drug: Novomix30

INTERVENTIONS:
Drug: Metformin — start with metformin，from 500mg bid,if metformin reach the biggest dosage，added gliclazide modified release tablets，afterthat，add acarbose
  Other Names: gliclazide modified release tablets; acarbose
  Arms: oral drugs
Drug: Lantus — started with insulin glargine 0.2 u/kg subcutaneous injection ，add dosage if glucose dose not reach the target.after that,you can add oral drugs（like oral drug group）
  Other Names: Metformin; gliclazide modified release tablets; acarbose
  Arms: lantus
Drug: Novomix30 — started with premixed insulin subcutaneous injection(0.4-0.6 u/kg divided into half before breakfast and dinner),and add dosage if glucose dose not reach the target.after that,you can add oral drugs ,as Group Oral Drugs
  Other Names: Metformin; gliclazide modified release tablets; acarbose
  Arms: Novomix30

SUMMARY:
Diabetic retinopathy (DR) is an important cause of blindness.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is an important cause of blindness, and its development of an irreversible process. DR is not only the overall progress and the level of blood sugar, and blood glucose fluctuations more closely, is the key to a smooth hypoglycemic delay DR progression.Diabetes control and complication trail(DCCT) study shows that even though glycemic control was no significant difference in blood glucose fluctuations ,DR also have a significant difference. In this study, three different glucose-lowering program for: (A) a single oral anti-diabetic drugs, (B) basal insulin and oral anti-diabetic drugs, (C) premixed insulin and oral anti-diabetic drugs for comparison. Focus on the stability and the impact of these three programs hypoglycemic long-term prognosis of the DR, and thus affect the molecular mechanisms of DR-based exploration of glucose fluctuations, to optimize blood glucose solutions, lower blood sugar steady, slow progression of DR ultimate clinical purposes.

The multi-center study is to cooperate, enrolled 600 cases of type 2 diabetes, observe the effects of different solutions on blood sugar glucose fluctuations and retinopathy, a total of 5 years of follow-up. This will be the first at home and abroad to compare the incidence of hypoglycemic effect programs on DR large multi-center, randomized, controlled clinical studies, clinical practice will optimize the treatment of type 2 diabetes theoretical and evidence-based medicine.

ELIGIBILITY:
Inclusion Criteria:

1. aged 30-65;
2. diagnosed to be type 2 diabetes in accordance with the WHO diagnostic criteria in 1999 .
3. diabetes duration for 5 years or less;
4. the glycosylated hemoglobin (HbA1c) is higher than or equal to7.0% ;
5. body mass index (BMI) 20-35 kg/m2;
6. fluorescein fundus angiography (FFA) showed no diabetic retinopathy;
7. women of childbearing-age have birth control plan for 5 years plan;

Exclusion Criteria:

1. pregnant or lactating women;
2. diabetes autoantibodies (GAD) antibodies positive;
3. occurred state of diabetic ketoacidosis, diabetes, high permeability, diabetes lactic acidosis within a half years ;
4. aspartate aminotransferase (AST), alanine aminotransferase (ALT) 2.5 times higher than normal ceiling, and/or serum creatinine (Cr) or 133 umol/l (1.5 mg/dl);
5. hemoglobin disease history which can affect determination of HbA1c;
6. have received a coronary angioplasty, coronary artery stent implantation, coronary artery bypass surgery, there was myocardial infarction, unstable angina, and clinical significance of abnormal ecg, cerebrovascular accident, or transient ischemic attack.
7. psychiatric patients;
8. any eye eyesight < 0.1 patients (WHO blind eye disease: keratitis, need serious cataract surgery, glaucoma, uveitis, high myopia shaft > 26.5 mm, history of ocular trauma;Other ophthalmology medical history: the central vein occlusion, branch vein occlusion, wet sex senile macular degeneration, etc.;
9. in eye surgery history, history of cataract surgery, and three months; Other serious diseases, the researchers think that don't fit into the patients

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2015-07; Primary Completion 2023-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of diabetic retinopathy | 5years
  5-year incidence rate of diabetic retinopathy（%）

SECONDARY OUTCOMES:
cardiovascular events | 5 years
  myocardial infarction, angina,or cardiac insufficiency with other causes
renal failure | 5years
  use urinary protein excretion rate（%） evaluate clinical course of diabetic nephropathy
glucose fluctuation | every one year in 5years
  we use continuous glucose monitoring system（CGMS）,made by Medtronic company USA,and assess within-day blood glucose excursions,Daytime blood sugar stability and the stability of postprandial blood glucose,including Standard Deviation Of Blood Glucose（SDBG）in mmol/L, largest amplitude of glycemic excursions(LAGE)in mmol/L, mean amplitude of glycemic excursions(MAGE) in mmol/L,low glycemic index(LBMI),coefficient variation fasting glucose parameters,Mean Of Daily Differences(MODD)in mmol/L.
oxidative stress | every one year in 5 years
  Glyoxalase 1(GLO-1)in pg/ml,Advanced glycation end products(AGEs）in pg/ml,Soluble Receptor for advanced glycation end products(sRAGE）in pg/ml.

OTHER OUTCOMES:
Metabolic indices | every three months in 5 years
  Fasting blood glucose（FBG）in mmol/L, postprandial blood glucose（PBG）in mmol/L, glycosylated hemoglobin（GHbA1c）in percentage.total cholesterol（TC), low density lipoprotein(LDL) and high density lipoprotein(HDL)in mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Mu panwei, Doctor, Principal Investigator — Employ
Locations (1):
- the third affiliated hospital of Sun yet-san university, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Klein BE. Overview of epidemiologic studies of diabetic retinopathy. Ophthalmic Epidemiol. 2007 Jul-Aug;14(4):179-83. doi: 10.1080/09286580701396720. PMID 17896294
- [Result] Kempen JH, O'Colmain BJ, Leske MC, Haffner SM, Klein R, Moss SE, Taylor HR, Hamman RF; Eye Diseases Prevalence Research Group. The prevalence of diabetic retinopathy among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):552-63. doi: 10.1001/archopht.122.4.552. PMID 15078674
- [Result] Fischbacher CM, Bhopal R, Unwin N, Walker M, White M, Alberti KG. Maternal transmission of type 2 diabetes varies by ethnic group: cross-sectional survey of Europeans and South Asians. Diabetes Care. 2001 Sep;24(9):1685-6. doi: 10.2337/diacare.24.9.1685-a. No abstract available. PMID 11522720
- [Result] Muggeo M, Zoppini G, Bonora E, Brun E, Bonadonna RC, Moghetti P, Verlato G. Fasting plasma glucose variability predicts 10-year survival of type 2 diabetic patients: the Verona Diabetes Study. Diabetes Care. 2000 Jan;23(1):45-50. doi: 10.2337/diacare.23.1.45. PMID 10857967
- [Result] White NH, Sun W, Cleary PA, Danis RP, Davis MD, Hainsworth DP, Hubbard LD, Lachin JM, Nathan DM. Prolonged effect of intensive therapy on the risk of retinopathy complications in patients with type 1 diabetes mellitus: 10 years after the Diabetes Control and Complications Trial. Arch Ophthalmol. 2008 Dec;126(12):1707-15. doi: 10.1001/archopht.126.12.1707. PMID 19064853
- [Result] Lin SD, Wang JS, Hsu SR, Sheu WH, Tu ST, Lee IT, Su SL, Lin SY, Wang SY, Hsieh MC. The beneficial effect of alpha-glucosidase inhibitor on glucose variability compared with sulfonylurea in Taiwanese type 2 diabetic patients inadequately controlled with metformin: preliminary data. J Diabetes Complications. 2011 Sep-Oct;25(5):332-8. doi: 10.1016/j.jdiacomp.2011.06.004. Epub 2011 Aug 2. PMID 21813293
- [Result] Bao YQ, Zhou J, Zhou M, Cheng YJ, Lu W, Pan XP, Tang JL, Lu HJ, Jia WP. Glipizide controlled-release tablets, with or without acarbose, improve glycaemic variability in newly diagnosed Type 2 diabetes. Clin Exp Pharmacol Physiol. 2010 May;37(5-6):564-8. doi: 10.1111/j.1440-1681.2010.05361.x. Epub 2010 Jan 17. PMID 20082624
- [Result] Bott S, Tusek C, Jacobsen LV, Endahl L, Draeger E, Kapitza C, Heise T. Insulin detemir under steady-state conditions: no accumulation and constant metabolic effect over time with twice daily administration in subjects with Type 1 diabetes. Diabet Med. 2006 May;23(5):522-8. doi: 10.1111/j.1464-5491.2006.01839.x. PMID 16681561
- [Result] Mu P, Lu H, Zhang G, Chen Y, Fu J, Wang M, Shu J, Zeng L. Comparison of fasting capillary glucose variability between insulin glargine and NPH. Diabetes Res Clin Pract. 2011 Jan;91(1):e4-7. doi: 10.1016/j.diabres.2010.09.026. PMID 20970870
- [Derived] Li S, Tang X, Luo Y, Wu B, Huang Z, Li Z, Peng L, Ling Y, Zhu J, Zhong J, Liu J, Chen Y. Impact of long-term glucose variability on coronary atherosclerosis progression in patients with type 2 diabetes: a 2.3 year follow-up study. Cardiovasc Diabetol. 2020 Sep 25;19(1):146. doi: 10.1186/s12933-020-01126-0. PMID 32977802
- [Derived] Tang X, Zhong J, Zhang H, Luo Y, Liu X, Peng L, Zhang Y, Qian X, Jiang B, Liu J, Li S, Chen Y. Visit-to-visit fasting plasma glucose variability is an important risk factor for long-term changes in left cardiac structure and function in patients with type 2 diabetes. Cardiovasc Diabetol. 2019 Apr 16;18(1):50. doi: 10.1186/s12933-019-0854-9. PMID 30992008